CLINICAL TRIAL: NCT02097095
Title: Substudy of GSK Protocol TB-018: Collection and Storage of Biological Samples for Evaluation of Correlates of Tuberculosis
Brief Title: Substudy of Protocol TB-018 (NCT01755598): Collection and Storage of Biological Samples for Evaluation of Correlates of TB (C-041-972)
Status: Completed | Type: Observational
Sponsor: Aeras (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: C-041-972
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Tuberculosis
Keywords: Correlates of risk; TB; Tuberculosis; Sub-study; TB-018
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Specimens for this sub-study are collected from an interventional Phase 2 study (TB-018 see NCT 01755598) and later analyzed for correlates of risk to tuberculosis.
  PBMC/Plasma; Whole Blood cell count; Intracellular RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccine group: TB vaccine GSK 692342 (M72/AS01E) administered on study TB-018
- Placebo Comparator: Placebo administered on study TB-018

SUMMARY:
This is an independent optional sub-study parallel to TB-018 (NCT01755598) in which biological samples will be collected for future investigations on biological correlates, markers or prognostic factors for TB disease. Subjects who consent to enroll in TB-018, "A phase IIb, double-blind, randomised, placebo-controlled study to evaluate the efficacy, safety and immunogenicity of GSK Biologicals' candidate tuberculosis (TB) vaccine GSK 692342 (M72/AS01E) against TB disease, in healthy adults aged 18-50 years, living in a TB endemic region", (see NCT 01755598) will be asked to participate in this sub-study. Subjects enrolled in TB-018 who also consent to C-041-972 will be followed according to the TB-018 protocol but will have additional blood samples collected for the sub-study.

DETAILED DESCRIPTION:
Additional information in the protocol

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this sub-study, subjects must be enrolled in TB-018 and provide separate written informed consent for C-041-972. See NCT 01755598 for inclusion criteria into TB-018.

Exclusion criteria:

To be eligible for this sub-study, subjects must be enrolled in TB-018 and provide separate written informed consent for C-041-972. See NCT 01755598 for exclusion criteria into TB-018.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who have consented to participate in TB-018 will be approached for participation in this sub-study. Subjects who have consented to participate in TB-018 are not required to participate in this sub-study.
Sampling Method: Probability Sample
Enrollment: 3253 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Collect and store biological samples for future use to evaluate potential biological markers correlated to the risk for tuberculosis. | 36 months in parallel with main study TB-018 (NCT01755598).
  Additional blood samples will be collected from participants that have agreed to be in this sub-study of TB-018 (NCT01755598).

SECONDARY OUTCOMES:
Collect and store biological samples for future use to evaluate immune correlates of protection from tuberculosis in subjects vaccinated with GSK 692342 (M72/AS01E). | 36 months in parallel with main study TB-018 (NCT01755598).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Landry, MS, Study Director — Aeras

IPD SHARING:
Plan to Share IPD: No